CLINICAL TRIAL: NCT00491959
Title: Phase 1 Study of Oral Mucosal Epithelial Cell Sheets in Patients Suffering From Corneal Stem Cell Insufficiency or Symblepharon
Brief Title: The Application of Oral Mucosal Epithelial Cell Sheets Cultivated on Amino Membrane in Patients Suffering From Corneal Stem Cell Insufficiency or Symblepharon.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to unstalbe cell sheet quality. We didn't use this tech on patients.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200701043D
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Limbal Insufficiency; Symblepharon
Keywords: oral mucosa; limbal insufficiency; transplantation; cornea; ocular surface
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cultured oral mucosa cell sheet transplantation — Cultivated oral mucosal cell sheets will be transplanted on the denuded corneal surface or the scleral surface of the symblepharon area. Therapeutic contact lenses will be applied after surgery.
  Other Names: oral mucosal cell sheets; Therapeutic contact lenses

SUMMARY:
Since cultivated autologous oral mucosal epithelial sheets on amniotic membrane have been reported to have good clinical results in treating patients with ocular surface disorders in both human or animal studies, and such technique has not been used in our hospital, the main purpose of this study is to use these cell sheets to treat patients with severe surface disorders, which include limbal insufficiency induced corneal surface problem, and symblepharon caused by severe conjunctival epithelial insufficiency. We will first choose patients who meet the surgical criteria, and these patients need to receive dental examination three months before surgery. Two weeks before transplantation, the oral mucosa tissue will be obtained by a dentist and the oral mucosal epithelial cell sheets will be cultivated on amniotic membrane until reaching confluency and stratification. During the transplantation surgery, the abnormal fibrovascular tissues on the ocular surface will be removed. The areas of symblepharon will also be released. The cultivated oral mucosal cell sheets will be transplanted on the denuded corneal surface or the scleral surface of the symblepharon area. Therapeutic contact lenses will be applied after surgery. After operation, the patients will be admitted for about two weeks. After discharge, the patients need to receive regular follow up weekly during the first two months, followed by biweekly follow up until postoperative 6 months. Afterward, the patients need to receive monthly follow up until postoperative 2 years. During the follow up, the data of the patients' visual acuity, intraocular pressure, slit lamp biomicroscopic findings, and in vivo confocal microscopic data will be obtained. The project plans to start from July 1st 2007 until June 30th 2010. We plan to enroll totally 20 patients.

DETAILED DESCRIPTION:
Cultivated autologous oral mucosal epithelial sheets on amniotic membrane have been reported to have good clinical results in treating patients with ocular surface disorders in both human or animal studies, and such technique has not been used in our hospital, the main purpose of this study is to use these cell sheets to treat patients with severe surface disorders, which include limbal insufficiency induced corneal surface problem, and symblepharon caused by severe conjunctival epithelial insufficiency. We will first choose patients who meet the surgical criteria, and these patients need to receive dental examination three months before surgery. Two weeks before transplantation, the oral mucosa tissue will be obtained by a dentist and the oral mucosal epithelial cell sheets will be cultivated on amniotic membrane until reaching confluency and stratification. During the transplantation surgery, the abnormal fibrovascular tissues on the ocular surface will be removed. The areas of symblepharon will also be released. The cultivated oral mucosal cell sheets will be transplanted on the denuded corneal surface or the scleral surface of the symblepharon area. Therapeutic contact lenses will be applied after surgery. After operation, the patients will be admitted for about two weeks. After discharge, the patients need to receive regular follow up weekly during the first two months, followed by biweekly follow up until postoperative 6 months. Afterward, the patients need to receive monthly follow up until postoperative 2 years. During the follow up, the data of the patients' visual acuity, intraocular pressure, slit lamp biomicroscopic findings, and in vivo confocal microscopic data will be obtained. The project plans to start from July 1st 2007 until June 30th 2010. We plan to enroll totally 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with bilateral limbal insufficiency

Exclusion Criteria:

* ocular diseases other than limbal insufficiency glaucoma diseases of retina or optic nerve

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
condition of ocular surface | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Rong Hu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan